CLINICAL TRIAL: NCT05539521
Title: Efficacy and Safety of Remimazolam Besylate Versus Propofol for Sedation in Critically Ill Patients With Deep Sedation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaobo Yang, MD, MD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WUHICU202202
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Critically Ill; Deep Sedation
Keywords: Remimazolam besylate; Propofol; Intensive care unit; Deep sedation
MeSH Terms: conditions — Critical Illness | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Besylate (Experimental): Patients in the remimazolam group received remimazolam besylate at an initial infusion rate of 0.3 mg/kg/h and adjusted to maintain a Narcotrend index between 13 and 64.
  Interventions: Drug: Remimazolam Besylate
- Propofol (Active Comparator): Patients in the propofol group received propofol at an initial infusion rate of 3.0 mg/kg/h and adjusted to maintain a Narcotrend index between 13 and 64.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam Besylate — sedation drugs
  Arms: Remimazolam Besylate
Drug: Propofol — Propofol
  Arms: Propofol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of remimazolam besylate compared to propofol for sedation in critically ill patients with deep sedation.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, controlled study using remimazolam besylate and propofol for sedation in critically ill patients with deep sedation. Subjects are randomized to remimazolam group and propofol group in a 1:1 ratio. Remifentanil is administered as the analgesic. Efficacy and safety profiles of remimazolam besylate are to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years;
* Expected to require deep sedation ≥8 hours;
* Requirement for deep sedation (a Narcotrend index between 13 and 64).

Exclusion Criteria:

* Body mass index (BMI) <18 or >30 kg/m2;
* Acute severe neurological disorder and any other condition interfering with RASS assessment;
* Systolic blood pressure less than 90 mm Hg after appropriate intravenous volume replacement and continuous infusions of 2 vasopressors;
* Heart rate less than 50 beats/min;
* Second- or third-degree heart block in the absence of a pacemaker;
* Unstable angina;
* Acute myocardial infarction;
* Left ventricular ejection fraction less than 30%;
* Contraindicate or allergic to study drugs;
* Moribund state;
* Acute hepatitis or serious hepatic dysfunction (Child-Pugh class C);
* Chronic kidney disease with glomerular filtration rate (GFR) < 60 ml/min/1.73m2;
* Alcohol abuse;
* Myasthenia gravis;
* Expected to have a general anesthesia within 8 hours;
* Pregnancy or lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The percentage of time in the target sedation range without rescue sedation | From the beginning of using study sedatives until being discharged from our ICU, the sedation target was changed, 48 hours after enrollment, or dead, whichever came first
  The percentage of time in the target sedation range without rescue sedation

SECONDARY OUTCOMES:
Adverse events | From the beginning of using study sedatives until being discharged from our ICU, the sedation target was changed, 48 hours after enrollment, or dead, whichever came first
  Adverse events
7-day ventitlator free time | From start of study to 7 days
  7-day ventitlator free time
Extubation at day 7 | From start of study to 7 days
  Extubation at day 7
Length of ICU stay | From start of study to 28 days
  Length of ICU stay
28-day mortality | From start of study to 28 days
  28-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: You Shang, Professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China